CLINICAL TRIAL: NCT03253263
Title: A Phase 2b, Multicenter, Randomized, Open-label, Two-Arm Study to Evaluate the Clinical Efficacy and Safety of OHB-607 Compared to Standard Neonatal Care for the Prevention of Bronchopulmonary Dysplasia, the Most Common Cause of Chronic Lung Disease of Prematurity
Brief Title: A Clinical Efficacy and Safety Study of OHB-607 in Preventing Bronchopulmonary Dysplasia in Extremely Premature Infants
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHB Neonatology Ltd. (Industry)
Responsible Party: Sponsor
Organization: Oak Hill Bio Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OHB-607-202; 2018-001393-16 (EudraCT Number); jRCT2071200076 (Registry Identifier: jRCT)
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Lung Disease of Prematurity; Intraventricular Hemorrhage; Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Retinopathy of Prematurity | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OHB-607 (Experimental): Participants will receive continuous IV infusion of OHB-607 through from birth up to PMA 29 weeks +6 days.
  Interventions: Drug: OHB-607
- Standard Neonatal Care (No Intervention): Standard neonatal care alone will be provided.

INTERVENTIONS:
Drug: OHB-607 — Participants will receive intravenous infusion of OHB-607 from birth up to PMA 29 weeks + 6 days.
  Other Names: Mecasermin Rinfabate
  Arms: OHB-607

SUMMARY:
The purpose of this study is to determine if an investigational drug can prevent Bronchopulmonary Dysplasia, reducing the burden of chronic lung disease in extremely premature infants, as compared to extremely premature infants receiving standard neonatal care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consents and/or assents must be signed and dated by the participant's parent(s) prior to any study related procedures. The informed consent and any assents for underage parents must be approved by the IRB/IEC (in accordance with local regulations).
2. Written informed consents and/or assents must be signed and dated by the participant's birth mother prior to providing study-related information related to birth mother medical history, pregnancy and the birth of the participant. The informed consent and any assents for underage birth mothers must be approved by the IRB/IEC (in accordance with local regulations).
3. Subjects must be between 23 weeks +0 days and 27 weeks +6 days GA, inclusive.

Exclusion Criteria:

1. Detectable major (or severe) congenital malformation identified before randomization.
2. Known or suspected chromosomal abnormality, genetic disorder, or syndrome, identified before randomization, according to the investigator's opinion.
3. Hypoglycemia at Baseline (blood glucose less than (<) 45 milligrams per deciliter [mg/dL] or 2.5 milli moles per liter [mmol/L]) which persists in spite of glucose supplementation, to exclude severe congenital abnormalities of glucose metabolism.
4. Clinically significant neurological disease identified before randomization according to cranial ultrasound (hemorrhages confined to the germinal matrix are allowed) and investigator's opinion.
5. Any other condition or therapy that, in the investigator's opinion, may pose a risk to the participant or interfere with the participant's potential compliance with this protocol or interfere with interpretation of results.
6. Current or planned participation in a clinical study of another investigational study treatment, device, or procedure (participation in non-interventional studies is permitted on a case-by-case basis).
7. The participant or participant's parent(s) is/are unable to comply with the protocol or is unlikely to be available for long-term follow-up as determined by the investigator.
8. Birth mother with active COVID-19 infection at birth or a history of severe COVID-19 infection (requiring intensive care hospitalization) during pregnancy.
9. Birth mother with known HIV or hepatitis (B, C, or E) infection.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Reduction in the incidence of severe Bronchopulmonary Dysplasia (BPD) at 36 weeks (±3 days) Postmenstrual Age (PMA), or death at or before 36 weeks PMA, whichever comes first as compared to the SNC group. | Baseline through 36 weeks postmenstrual age (PMA)
  Severe BPD is defined by the modified NICHD severity grading

SECONDARY OUTCOMES:
Reducing the burden of Chronic Lung Disease, as indicated by a reduction in time to final weaning off of Respiratory Technology Support (RTS) through 12 months Corrected Age (CA), as compared to the SNC group. | Baseline through 12 months CA
  The final weaning off of RTS is defined as the 7th consecutive day that the subject is off RTS.
Reduction in the incidence of severe BPD at 36 weeks (±3 days) PMA, or death at or before 36 weeks PMA, whichever comes first as compared to the SNC group. | Time Frame: Baseline through 36 weeks postmenstrual age (PMA)
  Severe BPD is defined based on the classification according to Jensen et al., 2019
Occurrence of severe (Grade 3 and 4) intraventricular hemorrhage (IVH) before 40 weeks PMA, as assessed by cranial ultrasound as compared to the SNC group | Baseline through 40 weeks postmenstrual age (PMA)
  Severe IVH as classified according to the Volpe criteria
To assess the effect of OHB-607 on occurrence of severe retinopathy of prematurity (ROP) (Stage 3 and above) up to 40 weeks PMA as compared to the SNC group | Baseline through 40 weeks postmenstrual age (PMA)
To assess the effect of OHB-607 on chronic respiratory outcomes as measured by the Chronic Lung Disease Prematurity Severity Score (CLDPSS) as compared to the SNC group at 12 months CA. | Baseline until 12 months CA using CLDPSS
The effect of OHB-607 on neurodevelopment is measured by the Cognitive, Language and Motor Scales of the Bayley Scales of Infant and Toddler Development (BSID) III as compared to the SNC group at 24 months CA. | Time Frame: Determined by the separate BSID III scales at 24 months CA
Chronic respiratory morbidity outcomes at 24 months CA | 24 months CA
Incidence and severity of BPD | Baseline through 36 weeks postmenstrual age (PMA)
  BPD severity is defined by the modified NICHD severity grading
Jensen BPD grade at 36 weeks PMA (± 3 days), as classified according to Jensen et al., 2019. Incidence of all severity grades of BPD as assessed by Jensen et al., 2019 | 36 weeks weeks postmenstrual age (PMA) (± 3 days)
Incidence and severity of IVH | Baseline through 36 weeks postmenstrual age (PMA)
  Incidence of all grades of IVH as assessed by centrally read CUS and classified according to the Volpe criteria
Neurodevelopment outcomes | From 6 months CA through 24 months CA
  Neurodevelopmental impairment, Physical and cognitive development will be measured by ASQ®-3 administered at 12 and 24 months CA.
Incidence of Retinopathy of Prematurity (ROP) | Baseline through 40 weeks PMA
  ROP is classified according to the International Classification
Mortality from randomization through to 24 months CA | From birth through 24 months CA
  Mortality rates from randomization to initial hospital discharge and from initial discharge through 24 months CA.
Exposure-response relationship between measured IGF-1 and Bronchopulmonary Dysplasia (BPD) | Baseline through 36 weeks PMA
  Blood samples will be collected to measure IGF-1 and these measured values will be associated with the incidence and severity grade of BPD
Exposure-response relationship between measured IGF-1 and intraventricular hemorrhage (IVH) | Baseline through 40 weeks PMA
  Blood samples will be collected to measure IGF-1 and these measured values will be associated with the incidence and severity grade of IVH
Exposure-response relationship between measured IGF-1 and necrotizing enterocolitis (NEC) | Baseline through 40 weeks PMA
  Blood samples will be collected to measure IGF-1 and these measured values will be associated with the incidence and severity grade of NEC
Exposure-response relationship between measured IGF-1 and Retinopathy of Prematurity (ROP) | Baseline through 40 weeks PMA
  Blood samples will be collected to measure IGF-1 and these measured values will be associated with the incidence and severity grade of ROP
To assess the safety profile of OHB-607 as compared to the SNC group. | Baseline through 24 months CA
  Incidence, severity, and causality assessment of Adverse Events (AEs) and Serious Adverse Events (SAEs), including Fatal AEs as per the neonatal adverse event severity scale.

CONTACTS AND LOCATIONS:
Locations (66):
- United States (23):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital of Orange County, California City, California
  - LAC USC Medical Center, Los Angeles, California
  - Jackson Memorial Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Minnesota - Children's Hospital and Clinics - St. Paul, Saint Paul, Minnesota
  - Children's Minnesota - Children's Hospital and Clinics, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Rochester, Rochester, New York
  - Maria Fareri Children's Hospital, Valhalla, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina Children Hospital, Charleston, South Carolina
  - UVA Children's Hospital, Charlottesville, Virginia
  - Virginia Commonwealth University - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Australia (3):
  - Royal Hospital for Women, Randwick, New South Wales
  - Royal Women's Hospital, Parkville
  - Mater Misericordiae Limited, South Brisbane
- Canada (2):
  - Sainte Justine Hospital, Montreal, Quebec
  - Mount Sinai Hospital, Toronto
- Oulun Yliopistollinen Sairaala, Oulu, Finland
- France (2):
  - Hôpital Antoine Béclère, Clamart, Hauts-de-Seine
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (3):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Klinikum Nürnberg, Nuremberg
- Cork University Maternity Hospital, Cork, Wilton, Ireland
- Italy (6):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliera Di Padova, Padua, Veneto
  - Azienda Ospedaliero-Universitaria Careggi SOD Neonatologia e Terapia Intensiva Neonatale, Florence
  - Istituto Giannina Gaslini-Istituto Pediatrico di Ricovero e, Genova
  - Presidio Ospedaliero Di Treviso Ca' Foncello, Treviso
- Japan (7):
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Nagano Children's Hospital, Azumino, Nagano
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Showa Medical University Hospital, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Tokyo
  - Osaka Women's and Children's Hospital, Izumi, Ôsaka
- Netherlands (3):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Academisch Medisch Centrum Amsterdam, Amsterdam-Zuidoost, North Holland
  - Wilhelmina Children Hospital-University Medical Center Utrecht, Utrecht
- Portugal (4):
  - Hospital Garcia de Orta, Almada
  - Maternidade Alfredo da Costa, Lisbon
  - Centro Hospitalar Lisboa, Lisbon
  - Centro Materno Infantil do Norte - Centro Hospital Universitario do Porto, E.P.E., Porto
- Hospital General Universitario Dr. Balmis, Alicante, Spain
- Sweden (2):
  - Skanes Universitetssjukhus, Lund
  - Karolinska Solna, Stockholm
- United Kingdom (8):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Ashford and St. Peter's Hospitals NHS Trust - St. Peter's Hospital, Chertsey, Surrey
  - University of Cambridge, Cambridge
  - University Hospital Coventry, Coventry
  - Liverpool Women's Hospital - PPDS, Liverpool
  - University College London, London
  - Chelsea and Westminster NHS Trust, London
  - St. Mary's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared in order to minimize the risk that individual patients could be re-identified, given that there are limited numbers of study participants at each study site per year.

REFERENCES:
- [Background] Kramer BW, Abman S, Daly M, Jobe AH, Niklas V. Insulin-like growth factor-1 replacement therapy after extremely premature birth: An opportunity to optimize lifelong lung health by preserving the natural sequence of lung development. Paediatr Respir Rev. 2023 Dec;48:24-29. doi: 10.1016/j.prrv.2023.05.001. Epub 2023 May 6. PMID 37268507
- [Background] Ley D, Hallberg B, Hansen-Pupp I, Dani C, Ramenghi LA, Marlow N, Beardsall K, Bhatti F, Dunger D, Higginson JD, Mahaveer A, Mezu-Ndubuisi OJ, Reynolds P, Giannantonio C, van Weissenbruch M, Barton N, Tocoian A, Hamdani M, Jochim E, Mangili A, Chung JK, Turner MA, Smith LEH, Hellstrom A; study team. rhIGF-1/rhIGFBP-3 in Preterm Infants: A Phase 2 Randomized Controlled Trial. J Pediatr. 2019 Mar;206:56-65.e8. doi: 10.1016/j.jpeds.2018.10.033. Epub 2018 Nov 22. PMID 30471715
- [Derived] Hellstrom W, Hortensius LM, Lofqvist C, Hellgren G, Tataranno ML, Ley D, Benders MJNL, Hellstrom A, Bjorkman-Burtscher IM, Heckemann RA, Savman K. Postnatal serum IGF-1 levels associate with brain volumes at term in extremely preterm infants. Pediatr Res. 2023 Feb;93(3):666-674. doi: 10.1038/s41390-022-02134-4. Epub 2022 Jun 9. PMID 35681088